CLINICAL TRIAL: NCT00795769
Title: Prevention of DMSO-Related Nausea and Vomiting by Prophylactic Administration of Ondansetron for Patients Receiving Autologous Cryopreserved Peripheral Blood Stem Cells
Brief Title: Ondansetron in Preventing Nausea and Vomiting in Patients Undergoing Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Principal Investigator, Leona Holmberg, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2247.00; NCI-2010-00325 (Registry Identifier: National Cancer Institute)
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Atypical Chronic Myeloid Leukemia, BCR-ABL Negative; Blastic Phase Chronic Myelogenous Leukemia; Chronic Eosinophilic Leukemia; Chronic Myelomonocytic Leukemia; Chronic Neutrophilic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; de Novo Myelodysplastic Syndromes; Disseminated Neuroblastoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Poor Prognosis Metastatic Gestational Trophoblastic Tumor; Previously Treated Myelodysplastic Syndromes; Primary Myelofibrosis; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Malignant Testicular Germ Cell Tumor; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Neuroblastoma; Recurrent Ovarian Epithelial Cancer; Recurrent Ovarian Germ Cell Tumor; Recurrent Small Lymphocytic Lymphoma; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Splenic Marginal Zone Lymphoma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage II Ovarian Epithelial Cancer; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Malignant Testicular Germ Cell Tumor; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Multiple Myeloma; Stage III Ovarian Epithelial Cancer; Stage III Small Lymphocytic Lymphoma; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Breast Cancer; Stage IV Chronic Lymphocytic Leukemia; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Ovarian Epithelial Cancer; Stage IV Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Primary Myelofibrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Testicular Neoplasms; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Neuroblastoma; Carcinoma, Ovarian Epithelial; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Leukemia, Hairy Cell; Multiple Myeloma; Breast Neoplasms | interventions — Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ondansetron therapy (Experimental): Patients receive ondansetron IV once 30-60 minutes before undergoing autologous peripheral blood stem cell transplantation.
  Interventions: Drug: ondansetron; Other: survey administration; Procedure: management of therapy complications

INTERVENTIONS:
Drug: ondansetron — Given IV
  Other Names: GR 38032F; GR-C507/75; Zofran
Other: survey administration — Correlative studies
Procedure: management of therapy complications — Ondansetron IV
  Other Names: complications of therapy, management of

SUMMARY:
RATIONALE: Ondansetron may help lessen or prevent nausea and vomiting in patients undergoing stem cell transplant.

PURPOSE: This phase II trial is studying how well ondansetron works in preventing nausea and vomiting in patients undergoing stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To determine whether the incidence of nausea and vomiting related to administration of autologous hematopoetic stem cells cryopreserved in DMSO can be reduced by the use of a single dose of intravenous ondansetron prior to the stem cell infusion.

II. To determine the number of patients who experience nausea and vomiting.

OUTLINE: Patients receive ondansetron IV once 30-60 minutes before undergoing autologous peripheral blood stem cell transplantation.

ELIGIBILITY:
Inclusion

* Autologous PBSC transplant patient
* English-speaking
* Planned cryopreserved PBSC infusion at the SCCA outpatient clinic

Exclusion

* History of prior autologous transplant
* Non-English-speaking
* Planned cryopreserved PBSC infusion at the UWMC inpatient unit
* Infusion of cryopreserved PBSC that are thawed and washed to remove DMSO prior to infusion
* Allergy or adverse reaction to ondansetron

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-08-08 (Actual); Primary Completion 2009-06-09 (Actual); Study Completion 2009-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leona Holmberg, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ondansetron Therapy
Started | 49
Completed | 49
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Ondansteron Therapy: Patients receive ondansetron IV once 30-60 minutes before undergoing autologous peripheral blood stem cell transplantation.
  ondansetron: Given IV
  survey administration: Correlative studies
  management of therapy complications: Ondansetron IV
Arm/Group | Ondansteron Therapy
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: years] | 52 [27 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Rates of Nausea or Vomiting After Ondansetron (Compared to FHCRC Historical Rates)
Description: Nausea Multinational Association of Supportive Care in Cancer Antiemesis Tool™ (MAT). Increased MAT scores represent worse outcome (score 0-10). Vomiting represented as present or absent.
Time Frame: Baseline up to 120 minutes
Measure: Count of Participants; unit: Participants
Groups:
- Ondansetron Therapy: Patients receive 16mg ondansetron IV once 30-60 minutes before undergoing autologous peripheral blood stem cell transplantation.
  ondansetron: Given IV
  survey administration: Correlative studies
  management of therapy complications: Ondansetron IV
Arm/Group | Ondansetron Therapy
Number analyzed (Participants) | 49
Participants
  MAT score >2 on arrival and pre-ondansetron | 23
  Baseline MAT score >2 prior to first ASCT infusion | 9
  MAT score increases >2 by end of infusion | 12
  Number of patients that vomited | 9
Statistical Analysis 1: Comparison: Ondansetron Therapy; 18% n=9 of the patients vomited compared to the FHCRC historic rate of 28%. p=0.03. PMID: 21372706 reference for historical data at FHCRC; Test type: Superiority or Other; p = 0.03, t-test, 1 sided
Statistical Analysis 2: Comparison: Ondansetron Therapy; Twelve patients (24%) had a greater than two-point increase in MAT score for nausea from baseline by the end of their infusion. That rate compares to the FHCRC historic rate of 58% (p <0.0001). PMID: 21372706 reference for historical data at FHCRC; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 11 months between August 2008-June 2009
Groups:
- Ondansteron Therapy: Patients receive 16 mg ondansetron IV once 30-60 minutes before undergoing autologous peripheral blood stem cell transplantation.
  ondansetron: Given IV
  survey administration: Correlative studies
  management of therapy complications: Ondansetron IV
Arm/Group | Ondansteron Therapy
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 18/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ondansteron Therapy (N=49)
nausea (Gastrointestinal disorders) | 9 — post stem cell infusion
nausea and vomiting (Gastrointestinal disorders) | 3 — post stem cell infusion. Also had > two point increase from baseline on MAT nausea score
vomiting (Gastrointestinal disorders) | 6 — post stem cell infusion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes